CLINICAL TRIAL: NCT00290394
Title: Study of PPAR Gamma Agonist-Rosiglitazone in Normotensive Type 2 Diabetics With Ambulatory Blood Pressure Monitoring
Brief Title: Ambulatory Blood Pressure Reduction After Rosiglitazone Treatment In Normotensive Type 2 Diabetic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baskent University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KA03/181
Record Dates: First submitted 2006-02-09; First posted 2006-02-13 (Estimated); Last update posted 2006-02-13 (Estimated); Status verified 2004-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Blood Pressure,; rosiglitazone,Diabetes Mellitus, Type 2,
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

INTERVENTIONS:
Drug: rosiglitazone(drug), blood pressure lowering effect

SUMMARY:
The purpose of this study was to determine the effects of rosiglitazone in normotensive type 2 diabetic patients with regard to its blood-pressure-reducing effects.

DETAILED DESCRIPTION:
The first study to evaluate the effects of troglitazone on blood pressure in humans was published recently, which demonstrated a 5/4 mm Hg reduction in ambulatory blood pressure in 18 nondiabetic obese subjects after 12 weeks' treatment. Another study in 18 hypertensive subjects with diabetes mellitus showed an 18/12 mm Hg decline in office blood pressure after 8 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Blood pressure of patients were in normotensive limits according to the JNC VII
* Diabetes mellitus treated with oral antidiabetics or diet

Exclusion Criteria:

* Any known hypertension, coronary artery disease, congestive hearth failure, renal disease or liver disease
* Anti-hypertensive treatment

Ages: 49 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2004-03; Study Completion 2004-08

PRIMARY OUTCOMES:
Ambulatory blood pressure monitors used to determine the subjects blood pressure before and after the treatment. At the end of three months period wit rosiglitazone treatment diastolic blood pressure decreased.

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan B Tutuncu, MD, Study Director — Medical Doctor, Endocrynology
Locations (1):
- Baskent University Ankara Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Takano H, Komuro I. Roles of peroxisome proliferator-activated receptor gamma in cardiovascular disease. J Diabetes Complications. 2002 Jan-Feb;16(1):108-14. doi: 10.1016/s1056-8727(01)00203-3. PMID 11872377
- [Background] Walker AB, Naderali EK, Chattington PD, Buckingham RE, Williams G. Differential vasoactive effects of the insulin sensitizers rosiglitazone (BRL 49653) and troglitazone on human small arteries in vitro. Diabetes. 1998 May;47(5):810-4. doi: 10.2337/diabetes.47.5.810. PMID 9588454
- [Background] Fujishima S, Ohya Y, Nakamura Y, Onaka U, Abe I, Fujishima M. Troglitazone, an insulin sensitizer, increases forearm blood flow in humans. Am J Hypertens. 1998 Sep;11(9):1134-7. doi: 10.1016/s0895-7061(98)00130-7. PMID 9752901
- [Background] Chen S, Noguchi Y, Izumida T, Tatebe J, Katayama S. A comparison of the hypotensive and hypoglycaemic actions of an angiotensin converting enzyme inhibitor, an AT1a antagonist and troglitazone. J Hypertens. 1996 Nov;14(11):1325-30. doi: 10.1097/00004872-199611000-00011. PMID 8934361
- [Background] Saku K, Zhang B, Ohta T, Arakawa K. Troglitazone lowers blood pressure and enhances insulin sensitivity in Watanabe heritable hyperlipidemic rabbits. Am J Hypertens. 1997 Sep;10(9 Pt 1):1027-33. doi: 10.1016/s0895-7061(97)00160-x. PMID 9324109
- [Background] Nolan JJ, Ludvik B, Beerdsen P, Joyce M, Olefsky J. Improvement in glucose tolerance and insulin resistance in obese subjects treated with troglitazone. N Engl J Med. 1994 Nov 3;331(18):1188-93. doi: 10.1056/NEJM199411033311803. PMID 7935656